CLINICAL TRIAL: NCT05727956
Title: Salvage Surgeries for Splanchnic Artery Aneurysms After Failed Endovascular Therapies: Cases Series
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chun Chieh Yeh, Clinical Professor of General Surgery, China Medical University Hospital
Other Study IDs: CMUH110-REC1-182
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Failure in Endovascular Therapy; Splanchnic Aneurysm; Mass Effect; Surgery
Keywords: salvage surgery; failed endovascular therapy; giant aneurysm; mass effect; jaundice; surgery
MeSH Terms: conditions — Jaundice

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Aneurysmectomy — Complete aneurysmectomy with end-to-end anastomosis for the true aneurysm or partial aneurysmectomy with a direct repair.

SUMMARY:
A retrospective review was performed for consecutive patients (from 2019 to 2021) who underwent salvage surgeries following failed endovascular therapies for splanchnic artery aneurysms in a tertiary referral center. Salvage operations include total aneurysmectomy with vascular reconstruction and partial aneurysmectomy with directly closing bleeders from the intraluminal space of the aneurysms.

DETAILED DESCRIPTION:
Salvage surgery for splanchnic artery aneurysm after failed endovascular trials includes one of the following three strategies: (1) aneurysmectomy along with the involved organ if the aneurysm is located within the parenchyma of solid organs (2) aneurysmectomy with vascular reconstruction if the aneurysm outside the solid organ (3)partial aneurysmectomy with direct closing the feeding vessel orifice if the aneurysm occurs in the hostile abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent salvage surgeries following failed endovascular therapies for splanchnic artery aneurysms
* The aneurysms were diagnosed based on medical history and computed tomography (CT)

Exclusion Criteria:

* Patients only underwent endovascular therapies for artery aneurysms
* The aneurysms are not located at the splanchnic artery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received surgical salvages after failed endovascular therapies for splanchnic arterial aneurysms in a tertiary university hospital (China Medical University Hospital, Taichung, Taiwan) between 2019 and 2021.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Survival outcomes after surgical intervention | From surgical intervention to the latest follow-up date (i.e., 2023-Jan-20)
  Survival outcomes (i.e., overall survival and symptoms-free survival in months) after salvage surgery for the splanchnic aneurysms were collected based on chart reviewing and telephone calls.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Chieh Yeh, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Department of Surgery, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ATLS Subcommittee; American College of Surgeons' Committee on Trauma; International ATLS working group. Advanced trauma life support (ATLS(R)): the ninth edition. J Trauma Acute Care Surg. 2013 May;74(5):1363-6. doi: 10.1097/TA.0b013e31828b82f5. No abstract available. PMID 23609291
- [Background] Akbulut S, Otan E. Management of Giant Splenic Artery Aneurysm: Comprehensive Literature Review. Medicine (Baltimore). 2015 Jul;94(27):e1016. doi: 10.1097/MD.0000000000001016. PMID 26166071
- [Result] Pulli R, Dorigo W, Troisi N, Pratesi G, Innocenti AA, Pratesi C. Surgical treatment of visceral artery aneurysms: A 25-year experience. J Vasc Surg. 2008 Aug;48(2):334-42. doi: 10.1016/j.jvs.2008.03.043. PMID 18644480
- [Result] Tipaldi MA, Krokidis M, Orgera G, Pignatelli M, Ronconi E, Laurino F, Laghi A, Rossi M. Endovascular management of giant visceral artery aneurysms. Sci Rep. 2021 Jan 12;11(1):700. doi: 10.1038/s41598-020-80150-2. PMID 33436829
- [Result] Pasha SF, Gloviczki P, Stanson AW, Kamath PS. Splanchnic artery aneurysms. Mayo Clin Proc. 2007 Apr;82(4):472-9. doi: 10.4065/82.4.472. PMID 17418076
- [Result] Shukla AJ, Eid R, Fish L, Avgerinos E, Marone L, Makaroun M, Chaer RA. Contemporary outcomes of intact and ruptured visceral artery aneurysms. J Vasc Surg. 2015 Jun;61(6):1442-7. doi: 10.1016/j.jvs.2015.01.005. Epub 2015 Mar 7. PMID 25752692
- [Result] Chaer RA, Abularrage CJ, Coleman DM, Eslami MH, Kashyap VS, Rockman C, Murad MH. The Society for Vascular Surgery clinical practice guidelines on the management of visceral aneurysms. J Vasc Surg. 2020 Jul;72(1S):3S-39S. doi: 10.1016/j.jvs.2020.01.039. Epub 2020 Mar 20. PMID 32201007
- [Result] Tetreau R, Beji H, Henry L, Valette PJ, Pilleul F. Arterial splanchnic aneurysms: Presentation, treatment and outcome in 112 patients. Diagn Interv Imaging. 2016 Jan;97(1):81-90. doi: 10.1016/j.diii.2015.06.014. Epub 2015 Aug 17. PMID 26292616
- [Result] Spiliopoulos S, Sabharwal T, Karnabatidis D, Brountzos E, Katsanos K, Krokidis M, Gkoutzios P, Siablis D, Adam A. Endovascular treatment of visceral aneurysms and pseudoaneurysms: long-term outcomes from a multicenter European study. Cardiovasc Intervent Radiol. 2012 Dec;35(6):1315-25. doi: 10.1007/s00270-011-0312-x. Epub 2011 Dec 7. PMID 22146976
- [Result] Pang TC, Maher R, Gananadha S, Hugh TJ, Samra JS. Peripancreatic pseudoaneurysms: a management-based classification system. Surg Endosc. 2014 Jul;28(7):2027-38. doi: 10.1007/s00464-014-3434-9. Epub 2014 Feb 12. PMID 24519028
- [Result] Marone EM, Mascia D, Kahlberg A, Brioschi C, Tshomba Y, Chiesa R. Is open repair still the gold standard in visceral artery aneurysm management? Ann Vasc Surg. 2011 Oct;25(7):936-46. doi: 10.1016/j.avsg.2011.03.006. Epub 2011 May 28. PMID 21620671
- [Result] Barrionuevo P, Malas MB, Nejim B, Haddad A, Morrow A, Ponce O, Hasan B, Seisa M, Chaer R, Murad MH. A systematic review and meta-analysis of the management of visceral artery aneurysms. J Vasc Surg. 2020 Jul;72(1S):40S-45S. doi: 10.1016/j.jvs.2020.05.018. PMID 32553135
- [Result] Androulakakis Z, Paspatis G, Hatzidakis A, Kokkinaki M, Papanicolaou N, Grammatikakis I, Liapi D, Kandylakis S. Gastric outlet obstruction caused by a giant gastroduodenal artery aneurysm: a case report. Eur J Gastroenterol Hepatol. 2001 Jan;13(1):59-61. doi: 10.1097/00042737-200101000-00011. PMID 11204812
- [Result] Saftoiu A, Iordache S, Ciurea T, Dumitrescu D, Popescu M, Stoica Z. Pancreatic pseudoaneurysm of the superior mesenteric artery complicated with obstructive jaundice. A case report. JOP. 2005 Jan 13;6(1):29-35. PMID 15650282
- [Result] Chapman BM, Bolton JS, Gioe SM, Conway WC. Gastroduodenal Artery Pseudoaneurysm Causing Obstructive Jaundice. Ochsner J. 2021 Spring;21(1):104-107. doi: 10.31486/toj.19.0110. PMID 33828434
- [Result] Jesinger RA, Thoreson AA, Lamba R. Abdominal and pelvic aneurysms and pseudoaneurysms: imaging review with clinical, radiologic, and treatment correlation. Radiographics. 2013 May;33(3):E71-96. doi: 10.1148/rg.333115036. PMID 23674782
- [Result] Madhusudhan KS, Venkatesh HA, Gamanagatti S, Garg P, Srivastava DN. Interventional Radiology in the Management of Visceral Artery Pseudoaneurysms: A Review of Techniques and Embolic Materials. Korean J Radiol. 2016 May-Jun;17(3):351-63. doi: 10.3348/kjr.2016.17.3.351. Epub 2016 Apr 14. PMID 27134524
- [Result] Zabicki B, Limphaibool N, Holstad MJV, Juszkat R. Endovascular management of pancreatitis-related pseudoaneurysms: A review of techniques. PLoS One. 2018 Jan 29;13(1):e0191998. doi: 10.1371/journal.pone.0191998. eCollection 2018. PMID 29377944
- [Result] Lopera JE. Embolization in trauma: principles and techniques. Semin Intervent Radiol. 2010 Mar;27(1):14-28. doi: 10.1055/s-0030-1247885. PMID 21359011
- [Result] Alsafi A, Bicknell CD, Rudarakanchana N, Kashef E, Gibbs RG, Cheshire NJ, Jenkins MP, Hamady M. Endovascular treatment of thoracic aortic aneurysms with a short proximal landing zone using scalloped endografts. J Vasc Surg. 2014 Dec;60(6):1499-506. doi: 10.1016/j.jvs.2014.08.062. Epub 2014 Sep 26. PMID 25264365
- [Result] Leyon JJ, Littlehales T, Rangarajan B, Hoey ET, Ganeshan A. Endovascular embolization: review of currently available embolization agents. Curr Probl Diagn Radiol. 2014 Jan-Feb;43(1):35-53. doi: 10.1067/j.cpradiol.2013.10.003. PMID 24290201
- [Result] Zyromski NJ, Vieira C, Stecker M, Nakeeb A, Pitt HA, Lillemoe KD, Howard TJ. Improved outcomes in postoperative and pancreatitis-related visceral pseudoaneurysms. J Gastrointest Surg. 2007 Jan;11(1):50-5. doi: 10.1007/s11605-006-0038-2. PMID 17390186
- [Result] ten Broek RP, Issa Y, van Santbrink EJ, Bouvy ND, Kruitwagen RF, Jeekel J, Bakkum EA, Rovers MM, van Goor H. Burden of adhesions in abdominal and pelvic surgery: systematic review and met-analysis. BMJ. 2013 Oct 3;347:f5588. doi: 10.1136/bmj.f5588. PMID 24092941
- [Result] Biondetti P, Fumarola EM, Ierardi AM, Carrafiello G. Bleeding complications after pancreatic surgery: interventional radiology management. Gland Surg. 2019 Apr;8(2):150-163. doi: 10.21037/gs.2019.01.06. PMID 31183325
- [Result] Grego FG, Lepidi S, Ragazzi R, Iurilli V, Stramana R, Deriu GP. Visceral artery aneurysms: a single center experience. Cardiovasc Surg. 2003 Feb;11(1):19-25. doi: 10.1016/s0967-2109(02)00121-7. PMID 12543567
- [Result] Krupski WC, Selzman CH, Floridia R, Strecker PK, Nehler MR, Whitehill TA. Contemporary management of isolated iliac aneurysms. J Vasc Surg. 1998 Jul;28(1):1-11; discussion 11-3. doi: 10.1016/s0741-5214(98)70194-6. PMID 9685125
- [Result] Moini M, Rasouli MR, Rayatzadeh H, Sheikholeslami G. Management of femoral artery pseudo-aneurysms in Iran: a single centre report of 50 cases. Acta Chir Belg. 2008 Mar-Apr;108(2):226-30. doi: 10.1080/00015458.2008.11680208. PMID 18557148
- [Result] Haseen MA, Faizan M, Beg MH, Asif N, Khalid S. Femoral artery pseudoaneurysm following trivial trauma: a rare case scenario. Indian Journal of Thoracic and Cardiovascular Surgery. 2015;31(1):34-7
- [Result] Saltzberg SS, Maldonado TS, Lamparello PJ, Cayne NS, Nalbandian MM, Rosen RJ, Jacobowitz GR, Adelman MA, Gagne PJ, Riles TS, Rockman CB. Is endovascular therapy the preferred treatment for all visceral artery aneurysms? Ann Vasc Surg. 2005 Jul;19(4):507-15. doi: 10.1007/s10016-005-4725-3. PMID 15986089
- [Result] Tulsyan N, Kashyap VS, Greenberg RK, Sarac TP, Clair DG, Pierce G, Ouriel K. The endovascular management of visceral artery aneurysms and pseudoaneurysms. J Vasc Surg. 2007 Feb;45(2):276-83; discussion 283. doi: 10.1016/j.jvs.2006.10.049. PMID 17264002
- [Result] Hemp JH, Sabri SS. Endovascular management of visceral arterial aneurysms. Tech Vasc Interv Radiol. 2015 Mar;18(1):14-23. doi: 10.1053/j.tvir.2014.12.003. Epub 2014 Dec 29. PMID 25814199
- [Result] Bougle A, Harrois A, Duranteau J. Resuscitative strategies in traumatic hemorrhagic shock. Ann Intensive Care. 2013 Jan 12;3(1):1. doi: 10.1186/2110-5820-3-1. PMID 23311726
- [Result] Coccolini F, Montori G, Catena F, Kluger Y, Biffl W, Moore EE, Reva V, Bing C, Bala M, Fugazzola P, Bahouth H, Marzi I, Velmahos G, Ivatury R, Soreide K, Horer T, Ten Broek R, Pereira BM, Fraga GP, Inaba K, Kashuk J, Parry N, Masiakos PT, Mylonas KS, Kirkpatrick A, Abu-Zidan F, Gomes CA, Benatti SV, Naidoo N, Salvetti F, Maccatrozzo S, Agnoletti V, Gamberini E, Solaini L, Costanzo A, Celotti A, Tomasoni M, Khokha V, Arvieux C, Napolitano L, Handolin L, Pisano M, Magnone S, Spain DA, de Moya M, Davis KA, De Angelis N, Leppaniemi A, Ferrada P, Latifi R, Navarro DC, Otomo Y, Coimbra R, Maier RV, Moore F, Rizoli S, Sakakushev B, Galante JM, Chiara O, Cimbanassi S, Mefire AC, Weber D, Ceresoli M, Peitzman AB, Wehlie L, Sartelli M, Di Saverio S, Ansaloni L. Splenic trauma: WSES classification and guidelines for adult and pediatric patients. World J Emerg Surg. 2017 Aug 18;12:40. doi: 10.1186/s13017-017-0151-4. eCollection 2017. PMID 28828034
- [Result] Kossak J, Janik J, Debski J, Rytlewski R, Salacinski A. Pseudoaneurysm of the gastroduodenal artery as a cause of obstructive jaundice. Med Sci Monit. 2001 Jul-Aug;7(4):759-61. PMID 11433208
- [Result] Donmez H, Men S, Dilli A, Soylu SO, Hekimoglu B. Giant gastroduodenal artery pseudoaneurysm due to polyarteritis nodosa as a cause of obstructive jaundice: imaging findings and coil embolization results. Cardiovasc Intervent Radiol. 2005 Nov-Dec;28(6):850-3. doi: 10.1007/s00270-004-0313-0. No abstract available. PMID 16132389
- [Result] Hamid HKS, Suliman AEA, Spiliopoulos S, Zabicki B, Tetreau R, Piffaretti G, Tozzi M. Giant Splenic Artery Pseudoaneurysms: Two Case Reports and Cumulative Review of the Literature. Ann Vasc Surg. 2020 Apr;64:382-388. doi: 10.1016/j.avsg.2019.10.061. Epub 2019 Oct 30. PMID 31676381
- [Result] Blomley MJ, Jackson JE. Case report: a gastroduodenal artery pseudoaneurysm presenting with obstructive jaundice and treated by arterial embolization. Clin Radiol. 1994 Oct;49(10):715-8. doi: 10.1016/s0009-9260(05)82668-6. PMID 7794312
- [Result] Sachdev U, Baril DT, Ellozy SH, Lookstein RA, Silverberg D, Jacobs TS, Carroccio A, Teodorescu VJ, Marin ML. Management of aneurysms involving branches of the celiac and superior mesenteric arteries: a comparison of surgical and endovascular therapy. J Vasc Surg. 2006 Oct;44(4):718-24. doi: 10.1016/j.jvs.2006.06.027. PMID 17011997